CLINICAL TRIAL: NCT05364736
Title: An Interventional Study for the Effects of Highland Barley β-glucan on the Management of Hypertension and Cardiovascular Risk
Brief Title: Effect of Prebiotics on Blood Pressure Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020HBβG-H
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hypertension; Gastrointestinal Microbiome
Keywords: Hypertension; Gastrointestinal Microbiome; Prebiotics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Participants, investigators and care providers at the scene are all blinded to the allocation of treatment group. Data collected will be analyzed by another investigator who is blinded to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Highland barley β-glucan group (Experimental): Participants will be given oral liquids mainly containing highland barley β-glucan once daily for 12 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Dietary Supplement: Highland barley β-glucan dietary supplement
- Placebo group (Placebo Comparator): Participants will be given oral liquids mainly containing Corn starch once daily for 12 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Other: Placebo controls

INTERVENTIONS:
Dietary Supplement: Highland barley β-glucan dietary supplement — 100 mL oral liquid mainly containing highland barley β-glucan once daily for 12 weeks
  Arms: Highland barley β-glucan group
Other: Placebo controls — Placebo with a similar appearance and taste to highland barley β-glucan supplement
  Arms: Placebo group

SUMMARY:
This survey is designed to investigate the effect of highland barley β-glucan supplementation on the regulatory of blood pressure, gut microbiota and cardiovascular risk fators in subjects with hypertention.

DETAILED DESCRIPTION:
Highland barley β-glucan belongs to the group of prebiotics and has been found to be associated with multiple health benefits. However, its protective role in subjects with hypertension are remain unclear. This study aims to examine the effect of 12-week prebiotics supplementation on blood pressure management in subjects with hypertension. By understanding the mechanism by which prebiotics exert the beneficial effects, we can better control the rising prevalence of hypertension, which is a major risk factor for cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age:30-65 years old
2. Newly diagnosed hypertension did not use antihypertensive drugs OR Systolic blood pressure ≥140mmHg on the physical examination OR Diastolic blood pressure ≥90mmHg on the physical examination.
3. BMI≥18 kg/m2

Exclusion Criteria:

1. Receiving or have been treated with antihypertensive drugs.
2. Complications including cardiovascular and cerebrovascular diseases such as coronary heart disease and stroke.
3. Severe liver or renal insufficiency (alanine aminotransferase, aspartate aminotransferase or alkaline phosphatase is greater than 3 times the upper limit of normal OR GFR<30ml/min/1.73m2).
4. Autoimmune diseases or thyroid diseases.
5. Women who are pregnant, nursing, or prepare to give birth during the trail.
6. Malignant disease, infectious disease, inflammatory disease and advanced liver disease.
7. Mental or intellectual abnormalities, unable to sign informed consent.
8. Complications including chronic gastrointestinal disease; or suffered from acute gastrointestinal diseases within 1 months before screening visit.
9. Received antibiotics, probiotics within 3 months before screening visit or throughout the trail.
10. Major operations were performed within six months of screening visit, or will be made during the trial.
11. Alcohol abuse (alcohol intake>60g/d for male and alcohol intake>40g/d for female)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-17 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of systolic blood pressure | baseline and 12 weeks
  changes of systolic blood pressure
changes of diastolic blood pressure | baseline and 12 weeks
  changes of diastolic blood pressure
changes of gut microbiota | baseline and 12 weeks
  changes of gut microbiota by metagenomics

SECONDARY OUTCOMES:
gut microbiota | baseline and 12 weeks
  changes of gut microbiota by metagenomics
pulse wave velocity | baseline and 12 weeks
  changes of pulse wave velocity by VP-1000plus from Omron
ankle Brachial Index | baseline and 12 weeks
  changes of ankle Brachial Index by VP-1000plus from Omron
microbial metabolite | baseline and 12 weeks
  changes of microbial metabolite by untargeted metabolomics
central aortic pressure | baseline and 12 weeks
  changes of central aortic pressure by VICORDER Complete Vascular Laboratory
flow-mediated dilation | baseline and 12 weeks
  changes of flow-mediated dilation by VICORDER Complete Vascular Laboratory
carotid-femoral pulse wave velocity | baseline and 12 weeks
  changes of carotid-femoral pulse wave velocity by VICORDER Complete Vascular Laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No